CLINICAL TRIAL: NCT04989621
Title: Orelabrutinib Plus Rituximab Followed by Maintenance With Orelabrutinib for Relapsed and Refractory Follicular Lymphoma(RR FL) ：a Single Arm, Open Label, Multi-center Phase II Study
Brief Title: Orelabrutinib Plus Rituximab Followed by Maintenance With Orelabrutinib for Relapsed and Refractory Follicular Lymphoma(RR FL)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Qingqing Cai, Chief physician, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2021-144
Record Dates: First submitted 2021-07-29; First posted 2021-08-04 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Follicular Lymphoma; Relapsed and Refractory Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular; Recurrence | interventions — orelabrutinib; Rituximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Orelabrutinib plus Rituximab followed by Maintenance with Orelabrutinib (Experimental): Induction therapy: Patients receive Orelabrutinib at a dose of 25 mg once daily on days 1-28 and rituximab at a dose of 375mg/m2 on day 1. Treatment cycles repeat every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  If patients achieve CR or PR or SD, they will be treated with maintenance therapy Maintenance therapy: Patients receive Orelabrutinib every day at a dose of 150mg for up to two years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Orelabrutinib and Rituximab; Drug: Orelabrutinib

INTERVENTIONS:
Drug: Orelabrutinib and Rituximab — Orelabrutinib 150mg po qd d1-28; Rituximab 375mg/m2 iv.drip d1.
  Other Names: induction treatment
Drug: Orelabrutinib — Orelabrutinib 150mg po qd

SUMMARY:
This phase 2 trial studies the efficacy and safety of orelabrutinib plus rituximab followed by maintenance with orelabrutinib for relapsed and refractory follicular lymphoma(RR FL)

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed grade 1, 2, or 3A FL;
* Patients received prior anti-lymphoma treatment;
* At least one evaluable lesion according to 2014 Lugano criteria;
* Age 18 years or older;
* Eastern Cooperative Oncology Group (ECOG) of 0-2;
* Life expectancy > 3 months;
* Able to participate in all required study procedures;
* Proper functioning of the major organs:

Exclusion Criteria:

* Patients who required warfarin or had a history of stroke or intracranial hemorrhage within 6 months, active transformed disease;
* Histological transformation of follicular lymphoma;
* Known central nervous system lymphoma;
* Received a prior allogeneic hematopoietic stem cell transplant. Prior autologous hematopoietic stem cell transplant is allowed;
* Subjects who have received prior treatment with ibrutinib, or other BTK inhibitors;
* Uncontrolled active infection, with the exception of tumor-related B symptom fever;
* Prior nitrosoureas within 6 weeks, chemotherapy within 3 weeks, therapeutic anticancer antibodies within 4 weeks, radio- or toxin-immunoconjugates within 10 weeks, radiation therapy or other investigational agents within 3 weeks, or major surgery within 4 weeks of first dose of study drug;
* Subjects who progressed or become refractory while on treatment with PI3K inhibitors are excluded. However, subjects who were responding to PI3K inhibitors, but had treatment discontinued due to toxicity, are eligible;
* Patients require treatment with strong CYP3A inhibitors;
* Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of Screening;
* Patients with active hepatitis B or active hepatitis C. Patients who are positive for hepatitis B Surface Antigen (HBsAg) or hepatitis C Virus (HCV) antibodies at screening stage must pass further detection of hepatitis B Virus (HBV) DNA (no more than 1000 IU/mL) and HCV RNA (no more than the lower limit of the detection method) in the row. Hepatitis B carriers, stable hepatitis B (DNA titer should not be higher than 1000 IU/mL) after drug treatment, and cured hepatitis C patients can be enrolled in the group;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Objective Response rate | 2 years
  Objective Response rate will be determined on the basis of investigator assessments according to 2014 Lugano criteria.

SECONDARY OUTCOMES:
Complete remission rate | 2 years
  Complete remission rate will be determined on the basis of investigator
Progression Free Survival | 4 years
  The time from the start of treatment to the progression of the tumor or death (due to any cause).
Overall Survival | 4 years
  The time from the start of treatment to time of death (due to any cause).
Duration of Response | 4 years
  The time from the first assessment of complete remission or partial remission to progressive disease or death (due to any cause).
Percentage of Participants With Adverse Events | 4 years
  Adverse Events will be determined and graded on the basis of investigator assessments according to NCI CTC AE 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Qingqing Cai, Study Director — Sun Yat-sen University
Locations (3):
- China (3):
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University,, Guangzhou, Guangdong
  - Sun Yat-sen Universitiy Cancer Center, Sun Yat-Sen University,, Guangzhou, Guangdong